CLINICAL TRIAL: NCT01890382
Title: Different Protein and Derivatives Supplementation Strategies Combined With Resistance Training in Pre-frail and Frail Elderly
Brief Title: Protein Intake and Resistance Training in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: The Pro Elderly Study
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Frail Elderly Syndrome
Keywords: resistance exercise; protein; creatine; leucine; aging
MeSH Terms: interventions — Whey Proteins; Whey; Creatine; Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control (Placebo Comparator): alanine as placebo to leucine (same dosage); corn starch as placebo to protein and/or creatine (same dosage)
  Interventions: Dietary Supplement: placebo
- whey protein (Experimental)
  Interventions: Dietary Supplement: Whey protein
- soy protein (Experimental)
  Interventions: Dietary Supplement: soy protein
- leucine supplementation (Experimental)
  Interventions: Dietary Supplement: leucine supplementation
- whey plus creatine (Experimental)
  Interventions: Dietary Supplement: whey plus creatine
- creatine (Experimental)
  Interventions: Dietary Supplement: creatine

INTERVENTIONS:
Dietary Supplement: Whey protein — 30 g in total; twice a day (morning and evening)
  Arms: whey protein
Dietary Supplement: whey plus creatine — whey protein combined with creatine (30 g and 6.0 g in total; twice a day, respectively)
  Arms: whey plus creatine
Dietary Supplement: leucine supplementation — 7.5 g/d in total; three times per day
  Arms: leucine supplementation
Dietary Supplement: soy protein — 30 g in total; twice a day
  Arms: soy protein
Dietary Supplement: creatine — 6.0 g in total; twice a day
  Arms: creatine
Dietary Supplement: placebo
  Arms: Control

SUMMARY:
Resistance training combined with protein or amino acids supplementation has been shown to be promising for mitigating age-related disabilities and comorbidities. Randomized controlled trials supporting this possibility are still scarce. These series of clinical trials aim to investigate the chronic effects of different strategies of protein and derivatives supplementation in association with resistance training on selected health-related parameters in pre-frail and frail elderly.This is a 16-month, double-blind, randomized, placebo-controlled, parallel-group clinical trial involving a series of investigations. Participants will be divided into nine groups, allowing the assessement of the effects of (1) isolated leucine supplementation; (2) protein source (whey vs. soy); (3) combination of whey protein and creatine; and (4) sexual dimorphism to the response of protein intake plus resistance training (men vs. women). All participants will undergo a supervised, resistance training program.

ELIGIBILITY:
Inclusion Criteria:

* elderly people
* frailty or pre-frailty, according to Fried et al., (2001) criteria.

Exclusion Criteria:

* on exogenous insulin and steroid-based drugs
* chronic obstructive pulmonary disease or respiratory failure
* use of protein and /or amine-based dietary supplements
* on restrictive diets (e.g. calorie or food group restrictions)
* on resistance training
* untreated cardiovascular, metabolic, or other chronic disease
* any musculoskeletal condition precluding resistance training

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
lean mass | 4 months
  assessed by Dual-energy X-ray absorptiometry
muscle function | 4 months
  assessed by a battery of physical tests

SECONDARY OUTCOMES:
bone mass | 4 months
  assessed by Dual-energy X-ray absorptiometry
insulin sensitivity | 4 months
  assessed by homeostasis model assessment (HOMA index)
health related-quality of life | 4 months
  assessed by Short-Form Health Survey (SF-36) (score range: 0 to 100, higher values mean better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Roschel H, Hayashi AP, Fernandes AL, Jambassi-Filho JC, Hevia-Larrain V, de Capitani M, Santana DA, Goncalves LS, de Sa-Pinto AL, Lima FR, Sapienza MT, Duarte AJS, Pereira RMR, Phillips SM, Gualano B. Supplement-based nutritional strategies to tackle frailty: A multifactorial, double-blind, randomized placebo-controlled trial. Clin Nutr. 2021 Aug;40(8):4849-4858. doi: 10.1016/j.clnu.2021.06.024. Epub 2021 Jul 3. PMID 34358827
- [Derived] Collins J, Longhurst G, Roschel H, Gualano B. Resistance Training and Co-supplementation with Creatine and Protein in Older Subjects with Frailty. J Frailty Aging. 2016;5(2):126-34. doi: 10.14283/jfa.2016.85. PMID 27224505